CLINICAL TRIAL: NCT05138822
Title: A Double-Blind, Double Dummy, Randomized, Phase 1b, Nitrofurantoin Controlled, Repeat Oral Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Microbiological Response of GSK3882347 in Female Participants With Acute Uncomplicated Urinary Tract Infection
Brief Title: Safety, Tolerability, Pharmacokinetic and Microbiological Investigation of GSK3882347 in Female Participants With Urinary Tract Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212943
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Uncomplicated Urinary Tract Infections; Urinary Tract Infections
Keywords: Microbiological response; Urinary tract infections (UTI); GSK3882347; Nitrofurantoin; Pharmacokinetics; Escherichia coli (E. coli)
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Intervention Model Description: This will be a randomized double-blind study and participants will be randomized to receive either GSK3882347 or nitrofurantoin in a 3:1 allocation ratio using an interactive response technology (IRT).
Who Masked: Participant, Investigator
Masking Description: This will be a randomized double-blind study with both participants and site staff blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GSK3882347 + Placebo (Experimental): Participants will be administered GSK3882347 plus placebo.
  Interventions: Drug: GSK3882347; Drug: Placebo
- Nitrofurantoin+ Placebo (Active Comparator): Participants will be administered nitrofurantoin plus placebo.
  Interventions: Drug: Nitrofurantoin; Drug: Placebo

INTERVENTIONS:
Drug: GSK3882347 — GSK3882347 will be administered on each dosing day.
  Arms: GSK3882347 + Placebo
Drug: Nitrofurantoin — Nitrofurantoin will be administered on each dosing day.
  Arms: Nitrofurantoin+ Placebo
Drug: Placebo — Placebo matching study drug (GSK3882347) or Nitrofurantoin will be administered on each dosing day.

SUMMARY:
This phase 1b study is a double-blind, double-dummy, nitrofurantoin-controlled study designed to evaluate microbiological response at the test of cure (ToC) visit along with safety, tolerability and pharmacokinetic (PK) response following daily oral dosing for 5 days of GSK3882347 in an adult female with uncomplicated urinary tract infections (uUTI). Comparator nitrofurantoin will be included in the study to ensure unbiased reporting of safety events. The study will be separated into 2 cohorts. Cohort 1 consists of an inpatient treatment period and PK analysis at frequent timepoints. Cohort 2 includes an outpatient treatment period and PK analysis conducted less frequently, at key trough timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to (>=)18 years of age and less than or equal to (<=)70 years
* The participant has 2 or more of the following clinical signs and symptoms of uncomplicated urinary tract infections (uUTI) with onset less than (<) 96 hours of the screening assessment: dysuria, frequency, urgency, or lower abdominal pain
* Participant has nitrite OR pyuria (≥ 10 white blood cells/ cubic millimeter [WBC/mm^3], OR > 5 WBC/high power field [HPF]) OR the presence of 2+ leukocyte esterase from a pre-treatment clean-catch midstream urine sample
* Participants with body mass index (BMI) >= 19.0 kilograms per square meter (kg/m^2)
* A female participant is eligible to participate who is not pregnant (as confirmed by a highly sensitive pregnancy test before the first dose of study intervention) or breastfeeding and one of the following conditions apply: 1) Woman participant of non-childbearing potential (WONCBP) Or 2) Woman participant of childbearing potential (WOCBP) using a contraceptive method that is highly effective, with a failure rate of < 1 percentage (%), during the study intervention period and up to 5 days post intervention
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* The participant has a BMI >= 40.0 kg/ m^2 or a BMI >=35.0 kg/ m^2 with obesity related health conditions such as high blood pressure or uncontrolled diabetes (non-fasting glucose value >300 milligram/deciliter [mg/dL])
* The participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of treatment failure and/or complications
* The participant has symptoms known or suspected to be caused by another disease process, such as asymptomatic bacteriuria, overactive bladder, chronic incontinence, or chronic interstitial cystitis
* The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction of the urinary tract, primary renal disease, or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract
* The participant has an indwelling catheter, nephrostomy, ureteral stent, or other foreign material in the urinary tract
* The participant who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptoms onset >=96 hours before the screening assessment, or a temperature >=101-degree Fahrenheit (°F) (>=38 degree Celsius [°C]), flank pain, chills, or any other manifestations suggestive of upper UTI
* The participant has anuria, oliguria, or significant impairment of renal function
* The participant presents at enrollment with a suspected sexually transmitted infection
* A positive confirmation of Coronavirus Disease 2019 (COVID-19) infection, or high clinical index of suspicion for COVID-19
* The participant has received treatment with other systemic antimicrobials or systemic antifungals within 1 week or 10 weeks for dalbavancin or oritavancin before study entry.
* Regular alcohol consumption within 6 months prior to the study with an average weekly intake of >14 units for females and one unit is equivalent to approximately 8 g of alcohol: a half-pint (250 mL) of beer, one glass (125 mL) of wine or one (35 mL) measure of spirits
* Unable to take nitrofurantoin. E.g. hypersensitivity to the active substance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — An adult female participant with 2 or more clinical signs and symptoms of acute urinary tract infections are included in this study activity.
Enrollment: 140 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Numbers of participants with microbiological response (responder/non-responder of GSK3882347) at the test of cure (TOC) visit | Day 10 to Day 13
  Microbiological response is defined as the response of less than (<)10^3 colony forming unit (CFU)/milliliter (mL) for all qualifying Escherichia coli (identified at baseline urine microbiology visit) at TOC visit, without receiving other systemic antimicrobials (rescue medications) prior to TOC

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 31
  AEs and SAEs will be collected.
Number of participants with clinically significant change from baseline in hematology parameters | Baseline (Day 1) and up to Day 31
  Blood samples will be collected for the assessment of hematology parameters.
Number of participants with clinically significant change from baseline in clinical chemistry | Baseline (Day 1) and up to Day 31
  Blood samples will be collected for the assessment of chemistry parameters.
Number of participants with clinically significant change from baseline in urinalysis | Baseline (Day 1) and up to Day 31
  Blood samples will be collected for the assessment of urinalysis parameters.
Number of participants with clinically significant change from baseline in vital signs | Baseline (Day 1) and up to Day 31
Number of participants with clinically significant change from baseline in 12- lead Electrocardiogram (ECG) findings | Baseline (Day 1) and up to Day 31
Plasma concentration of GSK3882347 single dose | Up to Day 5
  Blood samples will be collected for the concentrations of GSK3882347.
Urine concentration of GSK3882347 at 22-24-hour (h) interval collection post-dose | Up to Day 5
  Urine samples will be collected for the concentrations of GSK3882347.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (15):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Palmetto Bay, Florida
  - GSK Investigational Site, Sweetwater, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Smithfield, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Missouri City, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com